CLINICAL TRIAL: NCT06717061
Title: CAWA - Composed Abdominal Wall Analysis
Brief Title: Composed Abdominal Wall Analysis. Collecting Tissue and Blood From Patients Undergoing Elective Laparosopic Cholecystectomy. Objective to Describe the Normal Abdominal Wall
Acronym: CAWA
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Other Study IDs: RVasterbotten
Record Dates: First submitted 2024-08-19; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Hernia; Abdominal Wall
Keywords: hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma skin fascia muscle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Harvesting of study samples during planned intervention: Patients who are troubled by gallstone disease and are referred for laparoscopic surgery of the gallbladder at the surgical center Västerbotten in Skellefteå will receive oral and written information and will be asked to participate in the study.
  Once the blood samples have been taken, a research nurse will be on site in Skellefteå to collect the samples for centrifugation, pipetting and freezing. Serum and plasma will be shipped frozen to Umeå for analysis. Pieces of tissue are placed in formalin in the operating room and sent to the laboratory.
  Interventions: Procedure: Harvesting of biological material

INTERVENTIONS:
Procedure: Harvesting of biological material — During the sampling of biological material, the test subjects will be under general anesthesia, which is why the sampling will not mean increased pain or discomfort other than what is standard after a gallbladder operation with the peephole technique. . The sampling is not planned to be repeated, but is performed at the time when the patients perform their biliary surgery. During the sampling, centimeter-sized pieces of skin, fatty tissue, connective tissue and muscle are taken. Furthermore, serum and plasma will be collected. Two tubes of blood samples (10 ml total) are taken, centrifuged and pipetted before being frozen for later analysis. Pieces of tissue are placed in formalin before transport to the laboratory. The study form regarding the patient's basic state of health will be filled in by the operator on the day of surgery.

SUMMARY:
People who will be eligible to be asked about participation in the research project are individuals who seek planned care for surgery on their gallbladder due to gallstone disease. The group of patients is chosen as they can represent a normal material that enables comparison with hernia-specific disease in the abdominal wall.

Basic data such as height, weight, sex, age, medication and ASA class will be collected in the form of a study form and stored in a database in a pseudonymised form. During the sampling of biological material, the test subjects will be under general anesthesia, which is why the sampling will not mean increased pain or discomfort other than what is standard after a gallbladder operation with the minimally invasive technique. No additional wound area will be added to the test subjects as the sample pieces are taken from the area at the umbilicus where one operates by default. The sampling is not planned to be repeated, but is performed at the time when the patients perform their cholecystectomy. During the sampling, centimeter-sized pieces of skin, fatty tissue, connective tissue and muscle are taken. Furthermore, serum and plasma will be collected. Two tubes of blood samples (10 ml total) are taken, centrifuged and pipetted before being frozen for later analysis. Pieces of tissue are placed in formalin before transport to the laboratory. The study form regarding the patient's basic state of health will be filled in by the operator on the day of surgery and will be stored pseudonymized when the research subject is assigned a study number.

Patients who are troubled by gallstone disease and are referred for minimally invasive surgery of the gallbladder at the surgical center Västerbotten in Skellefteå will receive oral and written information and will be asked to participate in the study. Approximately 200 cholecystectomies are performed annually at Skellefteå hospital. We understand that within a reasonable period of time it will be possible to include 40 patients, which is the goal, also taking into account the exclusion criteria that exist. The inclusion of patients is expected to take approximately one year

ELIGIBILITY:
Inclusion Criteria:

- Individuals seeking planned care for surgery on their gallbladder due to gallstone disease

Exclusion Criteria:

* Disseminated cancer,
* Ongoing acute inflammation of the gallbladder,
* Known connective tissue disease,
* Cortisone medication,
* BMI >35,
* Clinically measured rectus diastasis of >4 cm and/or concurrent abdominal wall hernia
* Patients operated for abdominal wall hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who will be eligible to be asked about participation in the research project are individuals who seek planned care for surgery on their gallbladder due to gallstone disease. The group of patients is chosen as they can represent a normal material that enables comparison with hernia-specific disease in the abdominal wall
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Collagen composition differs between patients with abdominal wall hernia compared to patients without abdominal wall hernias | Five years from enrollment
  Are there detectable differences in collagen composition in the normal abdominal wall compared to patients who developed a primary or secondary abdominal wall hernia or abdominal rectus diastasis?

SECONDARY OUTCOMES:
Collagen turnover differs between patients with abdominal wall hernia compared to patients without abdominal wall hernias | Five years from enrollment.
  Are there detectable differences in hyaluronan levels, collagen metabolites, and other biological markers of collagen turnover in abdominal wall or blood when comparing patients with normal abdominal wall and subjects with diseased abdominal wall?

CONTACTS AND LOCATIONS:
Locations (1):
- Kirurgcentrum Västerbotten, Skellefteå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided